CLINICAL TRIAL: NCT03986593
Title: Cone-beam Computed Tomography Guided Percutaneous Cryoablation of Bone Metastases From Endocrine Tumors
Brief Title: Cryoablation of Bone Metastases From Endocrine Tumors
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study achieved n=17 participants (56.6% of the initial proposition) with a mean = 18 months follow-up. All patients completed 12 months follow-up or deceased. We chose to terminate and publish the data available.
Sponsor: Instituto do Cancer do Estado de São Paulo (Other)
Collaborators: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 990/2016
Record Dates: First submitted 2019-05-22; First posted 2019-06-14 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-05

CONDITIONS: Neoplasm Metastasis; Thyroid Neoplasm; Pheochromocytoma; Adrenal Neoplasm; Neuroendocrine Tumors; Bone Metastases
MeSH Terms: conditions — Neoplasm Metastasis; Thyroid Neoplasms; Pheochromocytoma; Adrenal Gland Neoplasms; Neuroendocrine Tumors | interventions — Cryosurgery

STUDY DESIGN:
Intervention Model Description: open, single-arm group, prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Cryoablation +- cementoplasty treated patients (Other): cone beam computed tomography guided cryoablation +- cementoplasty
  Interventions: Device: cryoablation

INTERVENTIONS:
Device: cryoablation — cryoablation of bone metastases by cone beam-CT image-guidance

SUMMARY:
This study will evaluate the clinical response and safety of cone beam computed-tomography guided percutaneous cryoablation in bone metastases from thyroid, adrenal and neuroendocrine tumors in 30 patients.

DETAILED DESCRIPTION:
Thyroid neoplasms, as well as adrenal and neuroendocrine tumors have the potential to metastasize to bone. About 3% of patients with well-differentiated thyroid carcinomas develop secondary bone lesions, while adrenal and neuroendocrine tumors have 10% and 13% bone metastases rates, respectively. Spinal metastases are associated to a worst prognosis. The progressive systemic disease, the post-operative complications, and the pre-operative neurologic impairment were associated to a worst global survival rate in the thyroid cancer. Additionally, extensive spinal instrumentation of metastatic thyroid carcinoma was associated to greater complication rates. Interventional radiology offers promising techniques for the minimally invasive approach of bone metastases. Image-guided percutaneous radiofrequency ablation and cryoablation techniques have been studied in clinical trials and are considered effective options in pain palliation of patients with bone metastatic disease. These techniques may be associated with conventional treatment, as well as radiation therapy and percutaneous embolization, avoiding major surgical interventions and its complications.

ELIGIBILITY:
Inclusion Criteria:

* patients with bone metastases from thyroid, adrenal or neuroendocrine tumor diagnosis, associated to one of the following: pain; risk fracture; risk of compression of spinal cord; hypercalcemia; performance status (ECOG) 0-3; mean life expectancy over one month;

Exclusion Criteria:

* age < 18 years
* active anticoagulant therapy or uncorrectable coagulopathy
* pregnancy or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2019-09-26 (Actual); Primary Completion 2022-10-15 (Actual); Study Completion 2023-05-29 (Actual)

PRIMARY OUTCOMES:
change in the local disease status of the cryoablation treated bone metastases | baseline (preprocedure); 01 week, 01 month, 03 months, 06 months, 12 months, 18 months, 24 months
  absence of neurological impairment and/or pain evaluated by clinical examination and brief pain inventory forms avoiding additional radiation therapy or surgery need

SECONDARY OUTCOMES:
evaluation of pain control | baseline (preprocedure); 01 week, 01 month, 03 months, 06 months, 12 months, 18 months, 24 months
  evaluation of pain control with the help of Brief Pain Inventory forms
evaluation of quality of life | baseline (preprocedure), 01 week, 01 month, 03 months, 06 months, 12 months, 18 months, 24 months
  evaluation of quality of life with the help of Brief Pain Inventory forms
number of participants with treatment-related adverse events according to CTCAE 5.0 | baseline (preprocedure); 01 week, 01 month, 03 months, 06 months, 12 months, 18 months, 24 months
  Major complications rates below 10%; Minor complication rates below 15%; Side effects rates bellow 20%; according to general guidelines (Society of Interventional Radiology - SIR);
imaging evaluation (CT or MRI) | baseline (preprocedure); 03 months, 06 months, 12 months, 24 months
  Computed tomography or Magnetic resonance imaging evaluation of eligible treated lesions
functional imaging evaluation (PET-CT) | baseline (preprocedure); immediate post-procedure; 06 months
  Computed tomography or Magnetic resonance imaging evaluation of eligible treated lesions

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo MC Freitas, PhD, Principal Investigator — Instituto do Cancer do Estado de São Paulo
Locations (1):
- Instituto do Cancer do Estado de São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available.
  Supporting information: Study protocol; Statistical Analysis Plan (SAP); Informed Consent Form (ICF); Clinical Study Report (CSR); Analytic Code; Time frame: Data will be available within 18 months of study completion. Access Criteria: Data access requests will be reviewed by an external Independent Review Panel. Requestors will be required to sign a Data Access Agreement.
Time Frame: Data will become available within 18 months of study completion and for 6 months.
Access Criteria: Data access requests will be reviewed by an external Independent Review Panel. Requestors will be required to sign a Data Access Agreement.

REFERENCES:
- [Background] de Freitas RM, de Menezes MR, Cerri GG, Gangi A. Sclerotic vertebral metastases: pain palliation using percutaneous image-guided cryoablation. Cardiovasc Intervent Radiol. 2011 Feb;34 Suppl 2:S294-9. doi: 10.1007/s00270-010-0085-7. Epub 2010 Dec 18. PMID 21170528
- [Background] Callstrom MR, Charboneau JW, Goetz MP, Rubin J, Wong GY, Sloan JA, Novotny PJ, Lewis BD, Welch TJ, Farrell MA, Maus TP, Lee RA, Reading CC, Petersen IA, Pickett DD. Painful metastases involving bone: feasibility of percutaneous CT- and US-guided radio-frequency ablation. Radiology. 2002 Jul;224(1):87-97. doi: 10.1148/radiol.2241011613. PMID 12091666
- [Background] Munk PL, Murphy KJ, Gangi A, Liu DM. Fire and ice: percutaneous ablative therapies and cement injection in management of metastatic disease of the spine. Semin Musculoskelet Radiol. 2011 Apr;15(2):125-34. doi: 10.1055/s-0031-1275595. Epub 2011 Apr 15. PMID 21500132
- [Background] Ferrer-Mileo L, Luque Blanco AI, Gonzalez-Barboteo J. Efficacy of Cryoablation to Control Cancer Pain: A Systematic Review. Pain Pract. 2018 Nov;18(8):1083-1098. doi: 10.1111/papr.12707. Epub 2018 Jun 7. PMID 29734509
- [Background] Callstrom MR, Dupuy DE, Solomon SB, Beres RA, Littrup PJ, Davis KW, Paz-Fumagalli R, Hoffman C, Atwell TD, Charboneau JW, Schmit GD, Goetz MP, Rubin J, Brown KJ, Novotny PJ, Sloan JA. Percutaneous image-guided cryoablation of painful metastases involving bone: multicenter trial. Cancer. 2013 Mar 1;119(5):1033-41. doi: 10.1002/cncr.27793. Epub 2012 Oct 12. PMID 23065947
- [Derived] de Freitas RMC, Hoff AO, Fragoso MCBV, Sousa AM, Danilovic DLS, de Castroneves LA, Grigio TR, Tsunemi MH, Buchpiguel CA, Caldas JGMP. Cryoablation of bone metastases in thyroid and adrenocortical cancers. Endocr Relat Cancer. 2026 Jan 30;33(1):e250306. doi: 10.1530/ERC-25-0306. Print 2026 Jan 1. PMID 41543023